CLINICAL TRIAL: NCT03997786
Title: A Multicenter, Randomized, Placebo and Active Comparator-controlled Clinical Trial to Study the Efficacy, Safety and Pharmacokinetics (PK) of Tildrakizumab in Pediatric Subjects From 6 to <18 Years of Age With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study of Tildrakizumab in Pediatric Subjects With Chronic Plaque Psoriasis
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TILD-19-12
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-09

CONDITIONS: Moderate-to-severe Chronic Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab; Etanercept

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will follow a two-component study design such that Part A will be an open label PK lead-in cohort of approximately 20 subjects. Part B will be a randomized trial component with approximately 100 subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (Active Comparator): Part A is a DOSE FINDING COMPONENT: OPEN LABEL PK lead-in and safety component
  Interventions: Drug: Tildrakizumab
- Part B Part 1: Placebo and active comparator controlled study (Experimental)
  Interventions: Drug: Placebo; Drug: Tildrakizumab; Drug: Etanercept
- Part B-1 and B-2: Randomized withdrawal and retreatment after relapse (Experimental)
  Interventions: Drug: Tildrakizumab; Drug: Placebo
- Part B 3: Efficacy and Safety Follow-up (No Intervention)
- Part C: LTE (Experimental)
  Interventions: Drug: Tildrakizumab

INTERVENTIONS:
Drug: Tildrakizumab — Week 0 (Day 1), Week 4 (Day 28) and week 16 (Day 112)
  Arms: Part A
Drug: Placebo — (Weeks 0 to 16)
  Arms: Part B Part 1: Placebo and active comparator controlled study
Drug: Tildrakizumab — (Weeks 16 to 52)
  Arms: Part B-1 and B-2: Randomized withdrawal and retreatment after relapse
Drug: Tildrakizumab — at every 12 weeks in open label fashion till 5 years (240 weeks).
  Arms: Part C: LTE
Drug: Tildrakizumab — (Weeks 0 to 16)
  Arms: Part B Part 1: Placebo and active comparator controlled study
Drug: Etanercept — (Weeks 0 to 16)
  Arms: Part B Part 1: Placebo and active comparator controlled study
Drug: Placebo — (Weeks 16 to 52)
  Arms: Part B-1 and B-2: Randomized withdrawal and retreatment after relapse

SUMMARY:
The study has been designed with three components. Part A is an open label PK study followed by a randomized trial component (Part B) followed by open label Long Term Extension (LTE).

The initial PK analysis is first done in adolescent subjects (12 to <18 years) before initiating the PK study in younger cohort (6 to <12 years)

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 6 to < 18 years of age, of either sex, of any race/ ethnicity, must weight greater than or equal to 15Kg.
* Diagnosis of predominantly plaque psoriasis for ≥6 months (as determined by subject interview and confirmation of diagnosis through physical examination by investigator).
* Moderate to severe psoriasis at baseline defined as: at least 10% Body Surface Area (BSA) involvement, PGA score ≥ 3, and PASI score ≥ 12
* Subject must be considered a candidate for systemic therapy, meaning psoriasis inadequately controlled by topical treatments (corticosteroids), and/or phototherapy, and/or previous systemic therapy
* Subject is considered to be eligible according to tuberculosis (TB) screening criteria
* A maximum of 2 QuantiFERON tests will be allowed. A re-test is only permitted if the first is indeterminate; the result of the second test will then be used.

Exclusion Criteria:

* Subject has predominantly non-plaque forms of psoriasis specifically erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new-onset guttate psoriasis
* Subject has laboratory abnormalities at screening including any of the following: Alanine transaminase (ALT) or aspartate transaminase, (AST) ≥2X the upper limit of normal, Creatinine ≥1.5X the upper limit of normal serum direct bilirubin ≥ 1.5 mg/dL, white blood cell count < 3.0 x 103/μL, and any other laboratory abnormality, which, in the opinion of the Investigator, will prevent the subject from completing the study or will interfere with the interpretation of the study results
* Subject who is expected to require topical therapy, phototherapy, or additional systemic therapy for psoriasis during the trial
* Female subjects of childbearing potential who are pregnant, intend to become pregnant (within 6 months of completing the trial), or are lactating. (Sexually active adolescent girls will be required to use contraception)
* Subject with presence of any infection or history of recurrent infection requiring treatment with systemic antibiotics within 2 weeks prior to Screening, or severe infection (e.g. pneumonia, cellulitis, bone or joint infections) requiring hospitalization or treatment with IV antibiotics within 8 weeks prior to Screening
* Positive human immunodeficiency virus (HIV) test result, hepatitis B surface (HBS) antigen, or hepatitis C virus (HCV) test result

Ages: 6 Years to 215 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2025-07-13 (Estimated); Study Completion 2031-12-05 (Estimated)

PRIMARY OUTCOMES:
Part A - Maximum Plasma Concentration | Day 3, 7 and 28 following first dose
Part A - Area under the plasma concentration-time curve | Day 3, 7 and 28 following first dose
Part A - Maximum Plasma Concentration | Weeks 4,8, and 12 following second dose
Part A - Area under the plasma concentration-time curve | Weeks 4,8, and 12 following second dose
Proportion of subjects with at least 75% improvement in the PASI response from baseline | Week 12
Proportion of subjects with PGA of "clear" or "almost clear" with at least a 2 grade reduction from baseline | Week 12
Number of subjects with adverse events | Week 52

SECONDARY OUTCOMES:
Proportion of subjects achieving Psoriasis Area & Severity Index (PASI) 50 from baseline | Week 12, 16, 28, 40, 52, 64, 76 and 88
Proportion of subjects achieving Psoriasis Area & Severity Index (PASI) 90 from baseline | Week 12, 16, 28, 40, 52, 64, 76 and 88
Proportion of subjects achieving Psoriasis Area & Severity Index (PASI) 100 from baseline | Week 12, 16, 28, 40, 52, 64, 76 and 88
Proportion of subjects achieving PASI 75 and PGA score of "clear" or "almost clear" with at least a 2 grade reduction from baseline | Week 16, 28, 40, 52, 64, 76 and 88
Change in quality of life as measured by Children's Dermatology Life Quality Index (CDLQI) | Week 108
  The CDLQI is a 10-item questionnaire that measures the impact of skin disease on children's (aged 2-15 years) quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The CDLQI total score was the sum of individual scores of question 1-10 and ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the children's life; 2-6 = small effect on the children's life; 7-12 = moderate effect on the children's life; 13-18 = very large effect on the children's life; 19-30 = extremely large effect on the children's life. Higher scores indicate more impact on quality of life of children.
Number of subjects with Adverse events | Week 108
Immunogenicity - Anti-drug antibody status | Week 108
Percent of subjects with severe infections | Week 108
  defined as any infection meeting the regulatory definition of a serious adverse event, or any infection requiring IV antibiotics whether or not reported as a serious event as per the regulatory definition
Percent of subjects with malignancies | Week 108
  including non-melanoma and melanoma skin cancer, but excluding carcinoma in situ of the cervix
Percent of subjects with confirmed major adverse cardiovascular events | Week 108
  major adverse cardiovascular events
Percent of subjects with drug- related hypersensitivity reactions | Week 108
  e.g. anaphylaxis, urticarial, angioedema, etc

OTHER OUTCOMES:
Relapse rates after withdrawal of treatment with tildrakizumab | Week 52
Rebound rates after withdrawal of treatment with tildrakizumab | Week 52
response to retreatment after relapse after withdrawal of treatment with tildrakizumab - Proportion of subjects with at least 75% improvement in the PASI response from baseline | Week 52
response to retreatment after relapse after withdrawal of treatment with tildrakizumab - Proportion of subjects with PGA of "clear" or "almost clear" with at least a 2 grade reduction from baseline | Week 52
Maintenance of response - Proportion of subjects with at least 75% improvement in the PASI response from baseline | Week 52
Maintenance of response - Proportion of subjects with PGA of "clear" or "almost clear" with at least a 2 grade reduction from baseline | Week 52

CONTACTS AND LOCATIONS:
Locations (50):
- United States (14):
  - Site 23, Birmingham, Alabama
  - Site 1, Fountain Valley, California
  - Site 2, Thousand Oaks, California
  - Site 4, Clearwater, Florida
  - Site 24, Coral Gables, Florida
  - Site 20, Miami, Florida
  - Site 7, Miami, Florida
  - Site 12, Orlando, Florida
  - Site 5, Bay City, Michigan
  - Site 16, Troy, Michigan
  - Site 22, Saint Joseph, Missouri
  - Site 8, Dallas, Texas
  - Site 10, South Jordan, Utah
  - Site 14, Spokane, Washington
- Hungary (5):
  - Site 63, Budapest
  - Site 62, Budapest
  - Site 61, Debrecen
  - Site 64, Kaposvár
  - Site 28, Szeged
- India (10):
  - Site 79, Ahmedabad
  - Site 70, Ahmedabad
  - Site 78, Chennai
  - Site 75, Kolkata
  - Site 76, Kolkata
  - Site 71, Lucknow
  - Site 73, Pune
  - Site 74, Surat
  - Site 77, Surat
  - Site 80, Warangal
- Poland (13):
  - Site 57, Bialystok
  - Site 55, Gdansk
  - Site 51, Katowice
  - Site 54, Lodz
  - Site 56, Lodz
  - Site 58, Lublin
  - Site 50, Ostrowiec Świętokrzyski
  - Site 59, Sosnowiec
  - Site 52, Szczecin
  - Site 53, Warsaw
  - Site 40, Wroclaw
  - Site 39, Wroclaw
  - Site 38, Wroclaw
- Slovakia (3):
  - Site 92, Bardejov
  - Site 91, Svidník
  - Site 90, Trnava
- Spain (5):
  - Site 41, Barcelona
  - Site 47, Las Palmas de Gran Canaria
  - Site 42, Madrid
  - Site 44, Valencia
  - Site 45, Valencia

IPD SHARING:
Plan to Share IPD: Undecided